CLINICAL TRIAL: NCT03729401
Title: Personalization of Long-Term Antiplatelet Therapy Using a Novel Combined Demographic/Pharmacogenomic Strategy - the RAPID EXTEND Randomized Study
Brief Title: Personalization of Long-Term Antiplatelet Therapy - RAPID EXTEND
Acronym: RAPID EXTEND
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Testing supplies unavailable.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180593
Record Dates: First submitted 2018-10-15; First posted 2018-11-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: 1-year post myocardial infarction; P2Y12 inhibitor; antiplatelet regimen
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Aspirin; Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DAPT - Aspirin and Ticagrelor (Active Comparator): As per results of the PEGASUS trial, patients will be treated with aspirin 81mg daily and ticagrelor 60mg twice daily
  Interventions: Drug: Active Comparator: Dual Antiplatelet Therapy (DAPT) - Aspirin 81 mg + Ticagrelor 60mg twice daily
- Ticagrelor Monotherapy (Experimental): Patients will only receive ticagrelor 60mg twice daily.
  Interventions: Drug: Ticagrelor Monotherapy: Ticagrelor 60 mg twice daily
- Personalized Therapy Arm (Experimental): Patients allocated to the personalized arm (PA) will have a DAPT score calculated. For those with a score of < 2, only aspirin at 81 mg daily will be prescribed. For those with a score of ≥ 2, P2Y12 inhibitor choice will be dependent on carrier status of CYP2C19 LOF alleles. Heterozygous or homozygous carriers will receive be prescribed ticagrelor 60mg twice daily and non-carriers with will be prescribed clopidogrel 75mg daily.
  Interventions: Drug: Personalized Therapy Arm: Aspirin 81 mg or Ticagrelor 60mg twice daily or Clopidogrel 75 mg once daily

INTERVENTIONS:
Drug: Active Comparator: Dual Antiplatelet Therapy (DAPT) - Aspirin 81 mg + Ticagrelor 60mg twice daily — DAPT with aspirin and ticagrelor
  Other Names: ASA, Brilinta
  Arms: DAPT - Aspirin and Ticagrelor
Drug: Ticagrelor Monotherapy: Ticagrelor 60 mg twice daily — Ticagrelor monotherapy
  Other Names: Brilinta
  Arms: Ticagrelor Monotherapy
Drug: Personalized Therapy Arm: Aspirin 81 mg or Ticagrelor 60mg twice daily or Clopidogrel 75 mg once daily — Personalized therapy based on risk score and genotyping
  Other Names: ASA, Brilinta, Plavix
  Arms: Personalized Therapy Arm

SUMMARY:
In patients after myocardial infarction (MI) (heart attacks) and treated with percutaneous coronary intervention (PCI), the current standard is dual antiplatelet therapy (DAPT), with aspirin and a P2Y12 receptor inhibitor, for 1 year of treatment. At 1 year, there are several options including: i) Ongoing DAPT (with aspirin and ticagrelor), ii) Selective treatment use of a P2Y12 inhibitor based on risk profiles.

This study is a pilot vanguard study to evaluate several strategies for choosing anti-platelet regimen among patients post MI and PCI at 1 year.

DETAILED DESCRIPTION:
The present study is a pilot/vanguard 3-arm study that seeks to compare 3 possible strategies for patients that are 1 year post MI and PCI. The 3 randomized groups include: i) aspirin and ticagrelor 60 mg twice daily, ii) monotherapy with ticagrelor 60 mg twice daily and iii) a personalized arm (PA), where patients will get selective therapy based on demographic and genetic risks.

The PA group will use a modified DAPT score based on patient demographics to decide whether P2Y12 treatment is warranted. For those patients where treatment is warranted, a bedside genetic test will be used to determine whether they are carriers of at-risk genotypes, which put them at risk for under-responsiveness to clopidogrel (one of the specific P2Y12 inhibitors). Those identified as carriers will be treated with ticagrelor while non-carriers will be treated with clopidogrel.

The study will act as a vanguard study to prove feasibility of enrollment and document overall bleeding rates. The long-term goal of the study is determine whether a personalized approach will decrease bleeding versus an approach of DAPT with ticagrelor and versus an approach with ticagrelor monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* >50 years old at 1-year after myocardial infarction (non-ST-elevation myocardial infarction (NSTEMI) or ST-elevation myocardial infarction (STEMI)) during which they had percutaneous coronary intervention (PCI)
* Compliant with dual antiplatelet therapy (DAPT) for ≥ 1 year without an ischemic or bleeding complication after PCI
* Still on DAPT regimen at enrollment
* Patients must have 1 of the following atherothrombotic risk enrichment criteria:

  i) Age≥ 65 years ii) Diabetes iii) 2nd Prior MI (>1 year ago) iv) multi-vessel coronary disease v) creatinine clearance (CrCl) <60 mL/min.

Exclusion Criteria:

* Intolerance to ticagrelor or clopidogrel
* >18 months post percutaneous coronary intervention (PCI) and myocardial infarction (MI)
* Requirement of a P2Y12 inhibitor
* Requirement of oral anticoagulation
* Take concurrent CYP3A inducing drugs which may interact with ticagrelor (e.g. anti-epileptic drugs)
* History of stroke, TIA or intracranial bleed
* Recent GI bleed or major surgery
* Life expectancy of < 1 year
* Platelet count < 100,000/μl
* Bleeding diathesis
* On dialysis
* Severe liver disease
* At risk for bradycardia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Bleeding Academic Research Consortium (BARC) Bleeding | 2 years post randomization
  BARC bleeding types 2,3 or 5
Feasibility for Patient Enrollment and Follow-up - measured by number of patients enrolled and followed over 2 years | 2 years
  Number of participants enrolled and followed: Target of 260 patients over 2 years with over 90% follow-up (Vanguard Study target)

SECONDARY OUTCOMES:
Thrombolysis in Myocardial Infarction (TIMI) bleeding | 1-3 years post randomization
  Incidence of TIMI bleeding - major and minor
Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) bleeding | 1-3 years post randomization
  Incidence of GUSTO bleeding - severe, moderate, mild
All Cause Mortality | 1 - 3 years post randomization
  Death due to any cause
Cardiovascular Mortality | 1 -3 years post randomization
  Death due to cardiovascular cause
Myocardial Infarction | 1 -3 years post randomization
  Myocardial infarction as defined by the 3rd universal definition on infarction
Stroke | 1-3 years
  Strokes defined as focal neurological deficit of >24 hrs and confirmed by imaging
Stent Thrombosis | 1 - 3 years post randomization
  Probable and definite stent thrombosis per ARC definition

CONTACTS AND LOCATIONS:
Overall Officials: Derek YF So, MD FRCPC, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonaca MP, Bhatt DL, Cohen M, Steg PG, Storey RF, Jensen EC, Magnani G, Bansilal S, Fish MP, Im K, Bengtsson O, Oude Ophuis T, Budaj A, Theroux P, Ruda M, Hamm C, Goto S, Spinar J, Nicolau JC, Kiss RG, Murphy SA, Wiviott SD, Held P, Braunwald E, Sabatine MS; PEGASUS-TIMI 54 Steering Committee and Investigators. Long-term use of ticagrelor in patients with prior myocardial infarction. N Engl J Med. 2015 May 7;372(19):1791-800. doi: 10.1056/NEJMoa1500857. Epub 2015 Mar 14. PMID 25773268
- [Background] Yeh RW, Secemsky EA, Kereiakes DJ, Normand SL, Gershlick AH, Cohen DJ, Spertus JA, Steg PG, Cutlip DE, Rinaldi MJ, Camenzind E, Wijns W, Apruzzese PK, Song Y, Massaro JM, Mauri L; DAPT Study Investigators. Development and Validation of a Prediction Rule for Benefit and Harm of Dual Antiplatelet Therapy Beyond 1 Year After Percutaneous Coronary Intervention. JAMA. 2016 Apr 26;315(16):1735-49. doi: 10.1001/jama.2016.3775. PMID 27022822
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention, 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery, 2012 ACC/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the Diagnosis and Management of Patients With Stable Ischemic Heart Disease, 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction, 2014 AHA/ACC Guideline for the Management of Patients With Non-ST-Elevation Acute Coronary Syndromes, and 2014 ACC/AHA Guideline on Perioperative Cardiovascular Evaluation and Management of Patients Undergoing Noncardiac Surgery. Circulation. 2016 Sep 6;134(10):e123-55. doi: 10.1161/CIR.0000000000000404. Epub 2016 Mar 29. No abstract available. PMID 27026020